CLINICAL TRIAL: NCT03109574
Title: A Pragmatic Multicenter Pilot Trial Evaluating the Cost-Effectiveness of BioFlo DuraMax Hemodialysis Catheter vs Standard of Care Catheter
Brief Title: Access in Dialysis for Better Outcomes in Patient Therapy
Acronym: ADOPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Osler Health System (Other)
Collaborators: Angiodynamics, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Sandra Donnelly, Clinical Nephrologist, William Osler Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: VA-BF410
Record Dates: First submitted 2017-03-20; First posted 2017-04-12 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Central Venous Catheter; Catheter-Related Bloodstream Infection (CRBSI) Nos
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care Device (Other): Current standard of care polyurethane catheter used at the hospital
  Interventions: Device: Standard of Care Catheter
- Study Device (Other): BioFlo DuraMax Chronic Hemodialysis Catheter
  Interventions: Device: BioFlo DuraMax Chronic Hemodialysis Catheter

INTERVENTIONS:
Device: BioFlo DuraMax Chronic Hemodialysis Catheter
  Arms: Study Device
Device: Standard of Care Catheter
  Arms: Standard of Care Device

SUMMARY:
This is a prospective, multi-center health economic study in Canada. Participants will be randomly assigned to receive either the study or control dialysis catheter. The primary objective is to evaluate resource utilization in Ontario related to hemodialysis catheter placement including tissue plasminogen activator (tPA) usage, catheter exchange rates, catheter patency, and missed dialysis days.

ELIGIBILITY:
Inclusion Criteria:

* Is indicated for a dialysis catheter for the purpose of attaining long-term vascular access for hemodialysis. Long-term vascular access is defined by physician anticipated duration of hemodialysis for three months or longer.
* Is ≥ 18 years of age.
* Is indicated to receive dialysis treatment at a location where dialysis treatment data will be accessible by the study team.
* Is able to comprehend and have signed the Informed Consent Form (ICF) to participate in the study.

Exclusion Criteria:

* Has known or suspected presence of other device-related infection, bacteremia, or septicemia or has been treated with antibiotics for documented or suspected infection within prior 45 days.
* Is receiving prophylactic anti-coagulation or anti-platelet pharmacotherapy for the purpose of central venous catheter (CVC) patency (anti-coagulation or anti-platelet pharmacotherapy for therapeutic indications do not exclude the patient from the study).
* Has severe chronic obstructive lung disease.
* Had past radiation therapy at the prospective insertion site.
* Had previous episodes of venous thrombosis or vascular surgical procedures at the prospective insertion site.
* Has local tissue factors that will prevent proper device stabilization and/or access.
* Has a stent placed in the vessel where the catheter will be placed
* Is pregnant
* History of drug or alcohol abuse in the past 12 months obtained from patient record and/or interview
* Subjects who weigh ≤ 30 kg.
* Has been previously enrolled in this clinical study, or is participating in another clinical study that is contraindicative to the treatment or outcomes of this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Resource utilization related to hemodialysis catheter placement - tPA | 1 year
  vials of tPA utilized (unit)

SECONDARY OUTCOMES:
Incidence of catheter-related complications | 1 year
  Includes thrombosis, infection, and any other catheter-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Donnelly, MD, Principal Investigator — William Osler Health System
Locations (3):
- Canada (3):
  - William Osler Health System, Brampton, Ontario
  - Halton Healthcare, Oakville, Ontario
  - Niagara Health System, Saint Catharines, Ontario